CLINICAL TRIAL: NCT01229800
Title: Efficacy, Safety and Tolerability of Split-dose of PEG Compared With NaP Solution for Colonoscopy Preparation: A Randomized, Controlled Trial
Acronym: SPEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Tae Oh Kim, Haeundae Paik Hospital, Inje University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HGI-2010-01
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-08

CONDITIONS: Bowel Preparation, Efficacy, Tolerability, Safety
Keywords: Polyethylene Glycol, Sodium Phosphate, Bowel preparation, Efficacy
MeSH Terms: interventions — Polyethylene Glycols; Solutions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Split dose PEG (Active Comparator): Group 1 (split-dose PEG regimen; Colyte, Taejoon Pharmaceuticals, Seoul, Korea; 236g PEG, 22.74g Na2SO4, 6.74g NaHCO3, 5.86g NaCl, and 2.97g KCl) ingested 2 liters of PEG at 6 PM on the day before the procedure and the remaining 2 liters in the early morning at least 2 hours prior to the procedure. Patients were instructed to take PEG 250 ml every ten minutes.
  Interventions: Drug: Polyethylene glycol
- Sodium phosphate(NaP) solution (Active Comparator): Group 2 (NaP regimen; Solin Oral, Korea Pharma., Seoul, Korea; 48g NaH2PO4 monosodium phosphate, 18g Na2HPO4 disodium phosphate) ingested 45ml NaP solution at 6 PM on the day before the procedure and remaining 45ml of NaP solution, separated temporally by minimum of 10 to 12 hours, at least 2 hours prior to the colonoscopy on the day of the procedure. Patients taking NaP solution were instructed to drink a minimum 1L of clear liquids during the evening on the day before the procedure and were encouraged to consume additional clear liquids.
  Interventions: Drug: Sodium phosphate(NaP) solution

INTERVENTIONS:
Drug: Polyethylene glycol — Group 1 (split-dose PEG regimen; Colyte, Taejoon Pharmaceuticals, Seoul, Korea; 236g PEG, 22.74g Na2SO4, 6.74g NaHCO3, 5.86g NaCl, and 2.97g KCl) ingested 2 liters of PEG at 6 PM on the day before the procedure and the remaining 2 liters in the early morning at least 2 hours prior to the procedure. Patients were instructed to take PEG 250 ml every ten minutes. Group 2 (NaP regimen; Solin Oral, Korea Pharma., Seoul, Korea; 48g NaH2PO4 monosodium phosphate, 18g Na2HPO4 disodium phosphate) ingested 45ml NaP solution at 6 PM on the day before the procedure and remaining 45ml of NaP solution, separated temporally by minimum of 10 to 12 hours, at least 2 hours prior to the colonoscopy on the day of the procedure.
  Other Names: Colyte(Taejoon Pharmaceuticals, Seoul, Korea)
  Arms: Split dose PEG
Drug: Sodium phosphate(NaP) solution — Group 2 (NaP regimen; Solin Oral, Korea Pharma., Seoul, Korea; 48g NaH2PO4 monosodium phosphate, 18g Na2HPO4 disodium phosphate) ingested 45ml NaP solution at 6 PM on the day before the procedure and remaining 45ml of NaP solution, separated temporally by minimum of 10 to 12 hours, at least 2 hours prior to the colonoscopy on the day of the procedure. Patients taking NaP solution were instructed to drink a minimum 1L of clear liquids during the evening on the day before the procedure and were encouraged to consume additional clear liquids.
  Other Names: Solin Oral (Korea Pharma., Seoul, Korea)
  Arms: Sodium phosphate(NaP) solution

SUMMARY:
: In several studies comparing of sodium phosphate solutions versus PEG, both regimen had similar efficacy of bowel cleansing and sodium phosphate solutions are more acceptable to patients because patient are required to consume smaller volume. But sodium phosphate solutions are associated with fluid and electrolyte disturbances, so use of sodium phosphate solution in routine medical check-up of outpatients is problematic. PEG can provide a rapid peroral approach to colon lavage without causing fluid and electrolyte disturbance. However, the need to ingest a large volume of fluid reduces patient compliance, and results in suboptimal bowel preparation. In order to overcome this disadvantage, several studies proved that split dose of PEG regimens were better quality preparation and more acceptable than single dose regimens. In Korea, need for outpatient or screening colonoscopy without laboratory test is increasing and split dose of PEG is used more frequently than other country in bowel preparation because of safety. But, superiority of split dose of PEG to sodium phosphate solution has not been demonstrated. The study was not yet existed about comparison of split dose PEG solution with sodium phosphate solution for bowel cleansing and tolerability in colonoscopy preparation. To use split dose of PEG in bowel preparation with medical evidence, we want to demonstrate split dose bowel preparation with PEG compared to sodium phosphate solutions provide a better colon cleansing efficacy and similar tolerability.

DETAILED DESCRIPTION:
Study design: Investigator-blinded, prospective, randomized controlled trial

Subjects

1. Entry criteria: Adult outpatients(at least 18 years of age, under 65 years) who undergo scheduled colonoscopy for screening, cancer surveillance or want procedure with/without non-specific gastrointestinal symptoms.
2. Exclusion criteria:

age under 18 years, elderly patients(>65 yrs), pregnancy, breast feeding, patient with bowel obstruction, and other structural intestinal disorders, gut hypomotility(chronic constipation(< 2 bowel movement/week for 1yr), hypomotility syndrome, megacolon, idiopathic pseudoobstruction), renal failure, congestive heart failure, liver failure, pre-existing electrolyte disturbance(hypercalcemia, hyperphosphatemia); refusal of consent to participate in the study.

Sampling design: Consecutive recruitment of consenting patients

Variables Predictor: split dose of PEG and sodium phosphate Primary Outcome: Quality of bowel preparation (Ottawa scale) Secondary Outcome: Tolerability (preparation completion, side effect) Confounding variables: age, gender, BMI, experience of colonoscopy, surgical history, bowel movement, comorbidity, indication, presence of GI symptoms, medication

Statistical issues

Hypothesis: Split dose bowel preparation with PEG will provide a better quality preparation and similar tolerability than that with sodium phosphate for morning colonoscopy.

Sample size.: Improving rate 20% in bowel cleansing efficacy(Ottawa scale), study power 80%, alpha-error(level of significance, P-value) 5%, mean value scale=5, effect size 1, SD=2.5-> sample size= 100/100

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients(at least 18 years of age, under 65 years) who undergo scheduled colonoscopy for screening, cancer surveillance or want procedure with/without non-specific gastrointestinal symptoms

Exclusion Criteria:

* age under 18 years, elderly patients(>,=65 yrs), pregnancy, breast feeding, patient with bowel obstruction, and other structural intestinal disorders, gut hypomotility(chronic constipation(< 2 bowel movement/week for 1yr), hypomotility syndrome, megacolon, idiopathic pseudoobstruction), renal failure, congestive heart failure, liver failure, pre-existing electrolyte disturbance(hypercalcemia, hyperphosphatemia); refusal of consent to participate in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 207 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of bowel preparation | Between August and October 2010.
  The primary end point of the study was to assess the quality of bowel preparation according to the Ottawa scale including cleanliness and fluid quantity.

SECONDARY OUTCOMES:
Safety and tolerability of bowel preparation | Between August and October 2010
  The secondary end points included patient tolerability and safety of bowel preparation using patient questionnaire consisted of compliance, acceptance, preference and adverse events such as abdominal pain and bloating, nausea and vomiting, headache and dizziness, sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Tae Oh Kim, M.D., PhD, Study Director — Inje University School of Medicine, Haeundae Paik Hospital; Eun Hee Seo, M.D., Principal Investigator — Inje University School of Medicine
Locations (1):
- Inje University School of Medicine, Haeundae Paik Hospital, Busan, South Korea

REFERENCES:
- [Derived] Seo EH, Kim TO, Kim TG, Joo HR, Park MJ, Park J, Park SH, Yang SY, Moon YS. Efficacy and tolerability of split-dose PEG compared with split-dose aqueous sodium phosphate for outpatient colonoscopy: a randomized, controlled trial. Dig Dis Sci. 2011 Oct;56(10):2963-71. doi: 10.1007/s10620-011-1772-1. Epub 2011 Jun 9. PMID 21656179